CLINICAL TRIAL: NCT00087802
Title: A Phase III Randomized Trial of Gemcitabine/Oxaliplatin (GEMOX) Versus Carboplatin/Paclitaxel (CP) as First-Line Therapy in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine/Oxaliplatin (GEMOX) vs Carboplatin/Paclitaxel (CP) in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9210; SR96669
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Oxaliplatin; CP protocol

ARMS (2):
- Stratum 1 (Active Comparator): Subjects will be randomized in a 1:1 allocation to either GEMOX or CP after signed consents and baseline evaluations are completed, allowing for safe entry into the study. In order to avoid an unbalanced distribution by baseline characteristics, randomization will be stratified by one factor: disease stage (in a 1:4 proportion for Stage IIIb vs. Stage IV or relapsed disease). Randomization schedules will be produced for each stratum, and treatment allocation will be carried out centrally
  Interventions: Drug: gemcitabine/Eloxatin (GEMOX)
- Stratum 2 (Active Comparator): Subjects will be randomized in a 1:1 allocation to either GEMOX or CP after signed consents and baseline evaluations are completed, allowing for safe entry into the study. In order to avoid an unbalanced distribution by baseline characteristics, randomization will be stratified by one factor: disease stage (in a 1:4 proportion for Stage IIIb vs. Stage IV or relapsed disease).
  Interventions: Drug: carboplatin/paclitaxel (CP)

INTERVENTIONS:
Drug: gemcitabine/Eloxatin (GEMOX) — GEMOX [gemcitabine/Eloxatin™ (Oxaliplatin) - 21 day cycle] Gemcitabine 1000 mg/m2 will be administered over 30 minutes on Days 1 and 8 and Eloxatin™ 130 mg/m2 will be administered over 2 hours on Day 1, after gemcitabine administration, every 21 days [3-week cycle]
  Arms: Stratum 1
Drug: carboplatin/paclitaxel (CP) — CP [carboplatin/paclitaxel - 21 day cycle]
  o Paclitaxel 225 mg/m2 will be administered over 3 hours on Day 1 followed by carboplatin at a dose calculated to produce an area under the concentration-time curve (AUC) of 6.0 over 30-60 minutes on Day 1 every 21 days [3-week cycle]
  Arms: Stratum 2

SUMMARY:
The purpose of this study is to compare combination treatment of gemcitabine + oxaliplatin (GEMOX) with carboplatin + paclitaxel (CP) to determine if there is a difference in response and safety between the two drug combinations for the treatment of advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, Stage IIIb or IV NSCLC, chemo or other systemic therapy naive
* One (1) unidimensionally measurable lesion
* ECOG Performance Status of 0 or 1, no peripheral neuropathy >Grade 1
* Patients with clinically stable brain metastases on a stable dose of (or no longer requiring) dexamethasone at registration will be eligible. Patients who have received cranial radiation for brain metastases must be at least 4 weeks from last radiation treatment.
* Recovery in full from any previous surgical procedure
* No history of an acute cardiac or CNS event within 6 months of entry or current clinical evidence of congestive heart failure or non-stable coronary artery disease

Exclusion Criteria:

* Hypersensitivity to any of the 4 study drugs
* Concurrent immunotherapy or participation in any investigational drug study within 4 weeks
* Serious uncontrolled intercurrent medical or psychiatric illness and organ allograft
* History of other malignancy within the last 5 years (except for squamous or basal cell carcinoma of the skin, carcinoma in situ of the cervix, or superficial transitional cell carcinoma of the bladder)
* Patient is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2004-03; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the relative efficacy, safety and clinical benefit of the GEMOX regimen compared to the standard combination regimen of CP as first-line treatment of Stage IIIB and IV NSCLC | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, MD, Study Director — Sanofi
Locations (69):
- United States (69):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Birmingham Hematology and Oncology Associates, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncology Associates - Hematology Oncology Physicians, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - South Florida Oncology & Hematology Consultants, Plantation, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Northwest Medical Specialists, PC, Niles, Illinois
  - Hematology Oncology Associates of Illinois, Skokie, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Oncology Associates of Cedar Rapids, Cedar Rapids, Iowa
  - Kansas City Oncology and Hematology Group, Overland Park, Kansas
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Arch Medical Services, Inc., St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, Latham, New York
  - New York Oncology Hematology, P.C., Rexford, New York
  - Interlakes Oncology & Hematology, P.C., Rochester, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - Piedmont Hematology Oncology Associates, PLLC., Winston-Salem, North Carolina
  - Dayton Oncology & Hematology, P.A., Kettering, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Texas Cancer Center - Abilene, Abilene, Texas
  - Texas Oncology, P.A., Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - Texas Cancer Center - Denton, Denton, Texas
  - El Paso Cancer Treatment Ctr-East, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - San Antonio Tumor and Blood Clinic, Fredericksburg, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Texas Oncology, P.A., Irving, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center - McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Hematology Oncology Associates of South Texas, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care and Research Center, Waco, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Fairfax Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Puget Sound Cancer Centers, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington